CLINICAL TRIAL: NCT04270747
Title: A Randomized, Double-masked, Phase 3 Study of ABP 938 Efficacy and Safety Compared to Aflibercept (Eylea®) in Subjects With Neovascular Age-related Macular Degeneration
Brief Title: A Study to Understand Effectiveness and Safety of ABP 938 Compared to Aflibercept (Eylea®) in Patients Suffering With Neovascular Age-related Macular Degeneration [Neovascular (Wet) AMD]
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20170542; 2019-002503-17 (EudraCT Number)
Record Dates: First submitted 2020-02-13; First posted 2020-02-17 (Actual); Results first posted 2024-01-05 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Neovascular (Wet) Age-related Macular Degeneration (AMD)
MeSH Terms: conditions — Macular Degeneration | interventions — aflibercept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: The study is double-masked; therefore, the investigators, study personnel, and the study subjects will remain masked to treatment allocation. Unmasking is only allowed in the case of an emergency, when knowledge of the investigational product is essential for the clinical management of the subject.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- ABP 938-Treatment Group A (Experimental): Subjects will receive 2 mg (0.05 mL) of ABP 938 by intravitreal (IVT) injection every 4 weeks for the first 3 doses (ie, baseline/day 1, week 4, and week 8) and every 8 weeks from week 16 until week 48.
  Interventions: Drug: ABP 938
- Aflibercept-Treatment Group B1 (Active Comparator): Subjects will receive 2 mg (0.05 mL) of aflibercept (Treatment Group B) by IVT injection every 4 weeks for the first 3 doses (ie, baseline/day 1, week 4, and week 8). Subjects will be re-randomized to receive aflibercept by IVT injection every 8 weeks from week 16 until week 48.
  Interventions: Drug: Aflibercept
- ABP 938-Treatment group B2 (Active Comparator): Subjects will receive 2 mg (0.05 mL) of aflibercept (Treatment Group B) by IVT injection every 4 weeks for the first 3 doses (ie, baseline/day 1, week 4, and week 8). Subjects will be re-randomized to receive ABP 938 by IVT injection every 8 weeks from week 16 until week 48
  Interventions: Drug: ABP 938; Drug: Aflibercept

INTERVENTIONS:
Drug: ABP 938 — Subject will receive ABP 938 2 mg (0.05 mL) IVT injection every 4 weeks for the first 3 doses, followed by once every 8 weeks
  Arms: ABP 938-Treatment Group A; ABP 938-Treatment group B2
Drug: Aflibercept — Subject will receive aflibercept 2 mg (0.05 mL) IVT injection every 4 weeks for the first 3 doses, followed by once every 8 weeks
  Other Names: Eylea®
  Arms: ABP 938-Treatment group B2; Aflibercept-Treatment Group B1

SUMMARY:
The purpose of this study is to compare the efficacy and safety of ABP 938 versus Aflibercept (Eylea®) in the treatment of neovascular age-related macular degeneration. Subjects will be randomized in a masked 1:1 ratio to receive 2 mg (0.05 mL) of either ABP 938 (Treatment Group A) or aflibercept (Treatment Group B) administered by intravitreal (IVT) injection.

DETAILED DESCRIPTION:
Approximately 566 subjects will be randomized in approximately 126 global sites.

This study consists of a screening period of up to 4 weeks, after which subjects will receive investigational product for 48 weeks, followed by a safety follow-up period to week 52, for a total study duration of up to 56 weeks.

Subjects will be randomized in a masked 1:1 ratio to receive 2 mg (0.05 mL) of either ABP 938 (Treatment Group A) or aflibercept (Treatment Group B) administered by IVT injection.

At week 8, subjects will be assessed for the primary endpoint. The primary endpoint is the change in Best Corrected Visual Acuity (BCVA) as measured by Early Treatment Diabetic Retinopathy Study (ETDRS) letter score from baseline to week 8, in order to assess the efficacy of ABP 938 compared to aflibercept.

Subjects will then be re-randomized at week 16 in a masked fashion such that:

* Subjects initially randomized to ABP 938 (Treatment Group A) will continue to receive ABP 938 by IVT injection every 8 weeks from week 16 until week 48
* Subjects initially randomized to aflibercept (Treatment Group B) will be re-randomized in a 1:1 ratio to either continue on aflibercept (Treatment Group B1) or transition to ABP 938 (Treatment Group B2) by IVT injection every 8 weeks from week 16 until week 48

ELIGIBILITY:
Inclusion Criteria:

* Subjects or their legally authorized representative must sign an Institutional Review Board/Independent Ethics Committee approved informed consent form before any study-specific procedures
* Men or women ≥ 50 years old
* Subjects must be diagnosed with neovascular (wet) AMD in the study eye
* Active treatment naïve subfoveal CNV lesions secondary to neovascular (wet) AMD including juxtafoveal lesions that affect the fovea as confirmed with SD OCT, FA and/or Fundus Photography (FP) in the study eye
* BCVA between 73 and 34 letters, inclusive, in the study eye using ETDRS testing
* Presence of intra and/or subretinal fluid as identified by SD-OCT attributable to active CNV in the study eye
* Central retinal thickness of > 270µm in the study eye as measured by the machine, calculated average thickness in the central 1 mm subfield (CST) by SD-OCT at screening

Exclusion Criteria:

Subjects are excluded if they meet any of the following criteria in the study eye:

* Total lesion size > 12 disc areas (30.5 mm^2, including blood, scars, and neovascularization) in the study eye
* Active CNV area (classic plus occult components) that is < 50% of the total lesion area in the study eye
* Scar, fibrosis, or atrophy involving the center of the fovea in the study eye
* Presence of retinal pigment epithelium tears or rips involving the macula in the study eye
* History of any vitreous hemorrhage within 4 weeks before randomization in the study eye
* Presence of other causes of CNV, including pathologic myopia (spherical equivalent of 8 diopters or more negative or axial length of 25 mm or more), ocular histoplasmosis syndrome, angioid streaks, choroidal rupture, or multifocal choroiditis in the study eye
* Prior vitrectomy or laser surgery of the macula (including photodynamic therapy or focal laser photocoagulation) in the study eye
* History of retinal detachment in the study eye
* Any history of macular hole of stage 2 and above in the study eye
* Any macular pathology that might limit vision i.e., Vitreomacular traction or significant epiretinal membrane in the study eye
* Any intraocular or periocular surgery within 3 months before randomization on the study eye, except lid surgery, which may not have taken place within 4 weeks before randomization, as long as it is unlikely to interfere with the injection
* Prior trabeculectomy or other filtration surgery in the study eye
* Uncontrolled glaucoma (defined as intraocular pressure ≥ 25 mmHg despite treatment with antiglaucoma medication) in the study eye
* Aphakia or pseudophakia with complete absence of posterior capsule (unless it occurred as a result of a yttrium aluminum garnet [YAG] posterior capsulotomy) in the study eye
* Previous therapeutic radiation in the region of the study eye
* History of corneal transplant or corneal dystrophy in the study eye
* Significant media opacities, including cataract, which might interfere with visual acuity or assessment of safety, in the study eye
* Any concurrent intraocular condition other than neovascular (wet) AMD in the study eye that, in the opinion of the investigator, requires planned medical or surgical intervention during the study or increases the risk to the subject beyond what is expected from standard procedures of intraocular injection, or which otherwise may interfere with the injection procedure or with evaluation of efficacy or safety

Subjects are excluded if they meet any of the following criteria in either eye:

* History or clinical evidence of uveitis, diabetic retinopathy, diabetic macular edema, or any other vascular disease affecting the retina, other than neovascular (wet) AMD
* Active intraocular inflammation or active or suspected ocular or periocular infection, within 2 weeks before randomization
* Active scleritis or episcleritis or presence of scleromalacia

Other Medical Conditions

• Active extraocular infection or history of extraocular infections as follows: A. any active infection for which systemic anti-infectives were used within 4 weeks before randomization B. recurrent or chronic infections or other active infection that, in the opinion of the investigator, might cause this study to be detrimental to the subject

* Acute coronary event or stroke within 3 months before randomization
* Uncontrolled, clinically significant systemic disease such as diabetes mellitus, hypertension, cardiovascular disease including moderate to severe heart failure (New York Heart Association class III/IV), renal disease, or liver disease
* Malignancy within 5 years EXCEPT treated and considered cured cutaneous squamous or basal cell carcinoma, in situ cervical cancer, OR in situ breast ductal carcinoma

Washouts and Nonpermitted Treatments

* Any prior ocular or systemic treatment, including another investigational product or surgery for neovascular (wet) AMD (including anti vascular endothelial growth factor [VEGF] therapy) in the study eye, except dietary supplements or vitamins
* Any ocular or systemic treatment including another investigational product or surgery for neovascular (wet) AMD (including anti VEGF therapy) in the fellow eye, within 30 days before randomization, except dietary supplements or vitamins
* Prior systemic anti-VEGF treatment as follows:
* Investigational or approved anti-VEGF therapy systemically within 3 months before randomization
* Aflibercept, ziv-aflibercept, or a biosimilar of aflibercept/ziv-aflibercept systemically at any time
* Any IVT therapy, including adrenocorticotropic hormone, in the study or fellow eye, or intramuscular or intravenous corticosteroids within 4 weeks before randomization. The use of long-acting steroids, either systemically or intraocularly, in the 3 months before randomization
* Currently receiving treatment with another investigational device or study drug, or less than 30 days or 5 half-lives (whichever is longer) since ending treatment on another investigational device or drug study(ies). Other investigational procedures while participating in this study are excluded

General

* For women: pregnant or breast feeding, or planning to become pregnant while enrolled in the study and for 3 months after the last dose of investigational product
* Sexually active subjects and their partners who are of childbearing potential (ie, neither surgically sterile nor postmenopausal) and not agreeing to use adequate contraception (eg, true abstinence, sterilization, birth control pills, Depo Provera injections, contraceptive implants, or other effective methods) while on study and for 3 months after the last dose of study drug. Male subjects must agree not to donate sperm during study and for 3 months following treatment with test article or until the scheduled end of the study (whichever is longer)
* Allergy or hypersensitivity to investigational product, to any of the excipients of ABP 938 or aflibercept, or to other study-related procedures/medications (eg, anesthesia, antiseptic, fluorescein dye)
* History or evidence of any other clinically significant disorder, condition, or disease (with the exception of those outlined above) that, in the opinion of the investigator or Amgen physician, if consulted, would pose a risk to subject safety or interfere with the study evaluation, procedures, or completion
* Subject likely to not be available to complete all protocol-required study visits or procedures, and/or to comply with all required study procedures (eg, Clinical Outcome Assessments) to the best of the subject and investigator's knowledge

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 576 (Actual)
Dates: Start 2020-06-22 (Actual); Primary Completion 2022-07-18 (Actual); Study Completion 2023-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (116):
- United States (40):
  - Associated Retina Consultants, Ltd. - Research, Phoenix, Arizona
  - Retina Consultants of Orange County, Fullerton, California
  - UCSD Shiley Eye Institute, Jacobs Retina Center, La Jolla, California
  - Jules Stein Eye Institute, UCLA, Los Angeles, California
  - Southern California Desert Retina Consultants, Palm Desert, California
  - Retina Consultants San Diego, Poway, California
  - Retina Consultants of Southern California, Redlands, California
  - Retinal Consultants Medical Group, Inc., Sacramento, California
  - Orange County Retina Medical Group, Santa Ana, California
  - Miramar Eye Specialists, Ventura, California
  - Colorado Retina Associates, Lakewood, Colorado
  - Retina Group of New England, Waterford, Connecticut
  - Florida Retina Consultants, Lakeland, Florida
  - Medeye Associates, Miami, Florida
  - Center for Retina and Macular Disease, Winter Haven, Florida
  - Southeast Retina Center, Augusta, Georgia
  - Georgia Retina, P.C., Marietta, Georgia
  - Retina Associates IL, Elmhurst, Illinois
  - Sabates Eye Center, Leawood, Kansas
  - Retina Associates New Orleans, Metairie, Louisiana
  - The Retina Care Center, Baltimore, Maryland
  - Specialty Eye Institute, Jackson, Michigan
  - Retina Center, Saint Louis Park, Minnesota
  - Retina Vitreous Surgeons of Central NY, PC, Liverpool, New York
  - Macula Care, New York, New York
  - Ophthalmic Consultants of the Capital Region - Ophthalmology, Troy, New York
  - Charlotte Eye Ear Nose & Throat Associates, P.A., Charlotte, North Carolina
  - Sterling Research Group, Cincinnati, Ohio
  - Eye Care Specialists, Kingston, Pennsylvania
  - Charleston Neuroscience Institute, Ladson, South Carolina
  - Black Hills Regional Eye Institute - Ophthalmology, Rapid City, South Dakota
  - Retina Research Institute of Texas, Abilene, Texas
  - Retina Consultants of Texas Research Centers, Bellaire, Texas
  - Texas Retina Associates, Dallas, Texas
  - Texas Retina Associates, Fort Worth, Texas
  - Ophthalmology Associates, Fort Worth, Texas
  - Premiere Retina Specialists, Midland, Texas
  - Retina Associates of South Texas, P.A., San Antonio, Texas
  - Retina Consultants of Houston, The Woodlands, Texas
  - Strategic Clinical Research, Willow Park, Texas
- Canada (2):
  - University of Ottawa Eye Institute, Ottawa, Ontario
  - Clinique d'ophtalmologie des laurentides, Boisbriand, Quebec
- Czechia (5):
  - Ocni klinika Pardubice, Pardubice
  - FN Kralovske Vinohrady, Prague
  - Vseobecna fakultni nemocnice v Praze, Prague
  - Axon Clinical, s.r.o., Prague
  - Krajska zdravotni, a.s. Masarykova nemocnice v Usti n/ Labem, Ústí nad Labem, Ústí Nad Labem
- Estonia (4):
  - East Tallinn Central Hospital - Eye Clinic, Tallinn, Harju
  - Eye Clinic of Dr. Krista Turman, Tallinn, Harju
  - Silmalaser OÜ, Tallinn, Harju
  - Eye Clinic of Tartu University Hospital, Tartu, Tartu
- Germany (7):
  - University Medical Center Freiburg, Freiburg im Breisgau, Baden-Wurttemberg
  - Klinikum Darmstadt, Darmstadt, Hesse
  - Universitätsmedizin Göttingen, Göttingen, Lower Saxony
  - St. Franziskus Hospital Münster, Münster, North Rhine-Westphalia
  - Universitätsmedizin Mainz, Mainz, Rhineland-Palatinate
  - Charité Universitätsmedizin Berlin KöR, Berlin
  - University Hospital Of Leipzig, Leipzig
- Hong Kong (2):
  - The University of Hong Kong - Department of Ophthalmology, Aberdeen
  - Prince of Wales Hospital - Department of Ophthalmology and Visual Sciences, Shatin, New Territories
- Hungary (8):
  - Ganglion Orvosi Központ, Pécs, Baranya
  - Szegedi Tudomanyegyetem Szent-Gyorgyi Albert Klinikai Kozpo, Szeged, Csongrád megye
  - Debreceni Egyetem Klinikai Központ, Debrecen, Hajdú-Bihar
  - Péterfy Kórház-Rendelintézet és Manninger Jen Országos Traumatológiai Intézet - Szemészeti Osztály, Budapest
  - Bajcsy-Zsilinszky Kórház és Rendelintézet, Budapest
  - Budapest Retina Intezet, Budapest
  - MH Egészségügyi Központ, Budapest
  - Semmelweis Egyetem, Budapest
- Israel (5):
  - Meir Medical Center, Kfar Saba, Central District
  - Soroka University Medical Center, Beersheba, Southern District
  - Bnai Zion Medical Center, Haifa, Southern District
  - Kaplan Medical Center, Rehovot
  - Assaf Harofeh Medical Center, Ẕerifin
- Italy (5):
  - Fondazione PTV Policlinico Tor Vergata, UNIT Patologie Retiniche, Rome, Lazio
  - UOC Oculistica Fondazione PU A.Gemelli IRCCS Un.Cattolica del Sacro Cuore, Rome, Lazio
  - Università degli Studi di Perugia, Ospedale Santa Maria della Misericordia, Clinica Oculistica, Perugia, Umbria
  - UO Oftalmologia Ciardella Pol. S.Orsola Malpighi AOU di Bologna, Bologna
  - "Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico, UO Oculistica Dipartimento di Chirurgia", Milan
- Japan (11):
  - Nagoya University Hospital, Nagoya, Aiti
  - Nagoya City University Hospital - Ophthalmology, Nagoya, Aiti
  - Asahikawa Medical University Hospital, Asahikawa, Hokkaidô
  - Fukushima Medical University Hospital - Ophthalmology, Fukushima, Hukusima
  - Kagoshima University Hospital - Ophthalmology, Kagoshima, Kagoshima-ken
  - Mie University Hospital, Tsu, Mie-ken
  - Nihon University Hospital - Ophthalmology, Tokyo, Tôkyô
  - University of Yamanashi Hospital, Chūō, Yamanashi
  - Akita University Hospital - Ophthalmology, Akita
  - Nagasaki University Hospital - Ophthalmology, Nagasaki
  - Kansai Medical University Hospital - Ophthalmology, Hirakata, Ôsaka
- Latvia (2):
  - P.Stradina Clinical University Hospital, Riga, Rga
  - Signes Ozolinas Doctor Praxis in Ophthalmology, Jelgava
- Lithuania (2):
  - Klaipedos Universitetine ligoniene, Klaipėda, Klaipdos Apskritis
  - Vilniaus Universiteto Ligonines Santariskiu Klinikos (VULSK), Vilnius, Vilnius County
- Mexico (3):
  - Asociación para Evitar la Ceguera en México I.A.P., México DF, Mexico City
  - Centro Medico Zambrano Hellion, Monterrey, Nuevo León
  - Centro de Retina Medica y Quirurgica S.C., Zapopan
- Poland (6):
  - Szpital Sw. Wojciecha, Poznan, Greater Poland Voivodeship
  - Profesorskie Centrum Okulistyki OKULISTYKA OPTIMUM, Gdansk, Pomeranian Voivodeship
  - Centrum Medyczne PROMED, Krakow
  - Centrum Diagnostyki i Mikrochirurgii Oka-Lens Sp. z o.o., Olsztyn
  - Centrum Medyczne UNO-MED, Tarnów
  - Klinika Okulistyczna "Jasne Blonia", Lodz, Ódzkie
- Clinical Center of Serbia, Belgrade, Serbia
- Slovakia (3):
  - Univerzitna nemocnica Bratislava, Bratislava, Bratislava Region
  - Fakultna nemocnica s poliklinikou Zilina, Žilina, Ilinský Kraj
  - Fakultna nemocnica Trencin, Trenčín, Treniansky Kraj
- South Korea (5):
  - Asan Medical Center, Seoul, Seoul Teugbyeolsi
  - Samsung Medical Center - Ophthalmology, Seoul, Seoul Teugbyeolsi
  - The Catholic University of Korea, Seoul St. Mary's Hospital - Neurology, Seoul, Seoul Teugbyeolsi
  - Seoul National University Hospital - Department of Ophthalmology, Seoul, Seoul Teugbyeolsi
  - Korea University Anam Hospital - Ophthalmology, Seoul
- Spain (5):
  - Hospital Universitario de Bellvitge, LHospitalet de Llobregat, Barcelona
  - Hospital Universitario Reina Sofía, Córdoba
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - FISABIO - Oftalmología Médica, Valencia

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 102 centers in Canada, Czech Republic, Estonia, Germany, Hong Kong, Hungary, Israel, Italy, Japan, South Korea, Latvia, Lithuania, Poland, Slovakia, Spain, and the United States between 22 June 2020 and 30 January 2023.
Pre-assignment Details: Both eyes were assessed at the screening visit for eligibility, and only 1 eye was selected from each participant as the study eye. If both eyes met the eligibility criteria, the study eye was the one with the worse best corrected visual acuity (BCVA).
Groups:
- ABP 938 / ABP 938: Participants were randomized to receive 2 mg (0.05 mL) of ABP 938 by intravitreal (IVT) injection in the study eye every 4 weeks for the first 3 doses (i.e., Baseline/Day 1, Week 4, and Week 8) and remained on ABP 938 dosing every 8 weeks from Week 16 until Week 48.
- Aflibercept / Aflibercept: Participants were randomized to receive 2 mg (0.05 mL) of aflibercept by IVT injection in the study eye every 4 weeks for the first 3 doses (i.e., Baseline/Day 1, Week 4, and Week 8) and were re-randomized to remain on aflibercept dosing every 8 weeks from Week 16 until Week 48.
- Aflibercept / ABP 938: Participants who were initially randomized to receive 2 mg (0.05 mL) of aflibercept by IVT injection in the study eye every 4 weeks for the first 3 doses (i.e., Baseline/Day 1, Week 4, and Week 8) were re-randomized to receive 2 mg (0.05 mL) of ABP 938 by IVT injection in the study eye every 8 weeks from Week 16 until Week 48.
Period: Through Week 16
Arm/Group | ABP 938 / ABP 938 | Aflibercept / Aflibercept | Aflibercept / ABP 938
Started | 288 | 288 | 0
Completed (Completed through Week 16) | 273 | 270 | 0
Not Completed | 15 | 18 | 0
Not completed — Adverse Event | 1 | 2 | 0
Not completed — Death | 0 | 2 | 0
Not completed — Consent Withdrawn | 3 | 3 | 0
Not completed — Physician Decision | 1 | 1 | 0
Not completed — Lost to Follow-up | 2 | 0 | 0
Not completed — Protocol Violation | 1 | 2 | 0
Not completed — Protocol Specified Criteria | 6 | 7 | 0
Not completed — Miscellaneous | 1 | 1 | 0
Period: Post Week 16
Arm/Group | ABP 938 / ABP 938 | Aflibercept / Aflibercept | Aflibercept / ABP 938
Started | 273 | 136 | 134
Received Treatment | 273 | 136 | 133
Completed | 251 | 125 | 123
Not Completed | 22 | 11 | 11
Not completed — Adverse Event | 7 | 5 | 1
Not completed — Death | 2 | 0 | 2
Not completed — Consent Withdrawn | 4 | 3 | 6
Not completed — Physician Decision | 3 | 1 | 1
Not completed — Lost to Follow-up | 2 | 1 | 0
Not completed — Requirement for Alternative Therapy | 1 | 0 | 0
Not completed — Requirement for Alternative Dosing Schedule | 2 | 1 | 0
Not completed — Miscellaneous | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set: Consisted of all randomized participants, with treatment as the randomized treatment regardless of actual treatment received. Participants were included in the treatment group in which they were initially randomized.
Groups:
- ABP 938: Participants were randomized to receive 2 mg (0.05 mL) of ABP 938 by IVT injection in the study eye every 4 weeks for the first 3 doses (i.e., Baseline/Day 1, Week 4, and Week 8) and remained on ABP 938 dosing every 8 weeks from Week 16 until Week 48.
- Aflibercept: Participants were randomized to receive 2 mg (0.05 mL) of aflibercept by IVT injection in the study eye every 4 weeks for the first 3 doses (i.e., Baseline/Day 1, Week 4, and Week 8) and were re-randomized to receive aflibercept or ABP 938 dosing every 8 weeks from Week 16 until Week 48.
- Total: Total of all reporting groups
Arm/Group | ABP 938 | Aflibercept | Total
Number analyzed (Participants) | 288 | 288 | 576
Age, Continuous [Mean (Standard Deviation); unit: Years] | 76.0 (7.93) | 76.0 (7.95) | 76.0 (7.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 151 | 171 | 322
  Male | 137 | 117 | 254
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 13 | 19
  Not Hispanic or Latino | 281 | 275 | 556
  Unknown or Not Reported | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 36 | 39 | 75
  Black or African American | 1 | 1 | 2
  Multiple | 1 | 0 | 1
  White | 250 | 248 | 498

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in BCVA at Week 8
Description: BCVA score was assessed based on the number of letters read correctly on the Early Treatment Diabetic Retinopathy Study (ETDRS) chart by the study eye at 4 meters. ETDRS letters score could range from 0 to 100 letters at each assessment.
  A positive change from Baseline in ETDRS letter score indicated an improvement in visual acuity in the study eye. Change from Baseline calculated as observed post-baseline value - Baseline value.
Time Frame: Baseline and Week 8
Population: Full Analysis Set: Consisted of all randomized participants, with treatment as the randomized treatment regardless of actual treatment received. Participants were included in the treatment group in which they were initially randomized. Analysis included participants with available data at Baseline and Week 8.
Measure: Mean (Standard Deviation); unit: Letters
Arm/Group | ABP 938 | Aflibercept
Number analyzed (Participants) | 279 | 281
Letters | 6.4 (8.18) | 6.5 (8.97)
Statistical Analysis 1: Comparison: ABP 938 vs Aflibercept; Difference in mean change from Baseline at Week 8; Test type: Other — A pre-specified similarity margin of (-3, 3) ETDRS letters was used to demonstrate clinical similarity for the mean change from Baseline in BCVA at Week 8; Difference between means = 0.1, 90% CI 2-sided [-1.1 to 1.3] — Estimated using analysis of covariance (ANCOVA) model adjusted for the stratification factors geographic region (East Asia, Europe, North America) and Baseline BCVA as covariates

2. Secondary Outcome: Percentage of Participants Who Maintained Vision at Week 52
Description: A participant was classified as maintaining vision if he/she lost fewer than 15 letters in ETDRS letter score, assessed in the study eye, compared to Baseline.
Time Frame: Week 52
Population: Full Analysis Set (Re-randomized): Consisted of all re-randomized participants, with treatment as the randomized treatment regardless of actual treatment received. Participants were included in the treatment group in which they were re-randomized. Analysis included participants with available data at Baseline and Week 52.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- ABP 938 / ABP 938: Participants who were initially randomized to receive 2 mg (0.05 mL) of ABP 938 by IVT injection in the study eye every 4 weeks for the first 3 doses (i.e., Baseline/Day 1, Week 4, and Week 8) and remained on ABP 938 dosing every 8 weeks from Week 16 until Week 48.
- Aflibercept / Aflibercept: Participants who were initially randomized to receive 2 mg (0.05 mL) of aflibercept by IVT injection in the study eye every 4 weeks for the first 3 doses (i.e., Baseline/Day 1, Week 4, and Week 8) and were re-randomized to remain on aflibercept dosing every 8 weeks from Week 16 until Week 48.
Arm/Group | ABP 938 / ABP 938 | Aflibercept / Aflibercept | Aflibercept / ABP 938
Number analyzed (Participants) | 251 | 125 | 123
Percentage of Participants | 95.6 [93.1 to 98.2] | 97.6 [94.9 to 100.0] | 95.9 [92.5 to 99.4]
Statistical Analysis 1: Comparison: ABP 938 / ABP 938 vs Aflibercept / Aflibercept; Risk difference in percentage of participants who maintained vision at Week 52; Test type: Other; Risk Difference (RD) = -2.1, 90% CI 2-sided [-5.2 to 2.2] — Estimated using the stratified Newcombe confidence limits (with Mantel-Haenszel weights) adjusting for stratification factors geographic region (East Asia, Europe, North America) and Baseline BCVA (BCVA < 64 letters, BCVA ≥ 64 letters)
Statistical Analysis 2: Comparison: Aflibercept / Aflibercept vs Aflibercept / ABP 938; Risk difference in percentage of participants who maintained vision at Week 52; Test type: Other; Risk Difference (RD) = -1.7, 90% CI 2-sided [-6.2 to 2.8] — [estimate comment as in outcome 2, analysis 1]

3. Secondary Outcome: Mean Change From Baseline in BCVA
Description: BCVA score was assessed based on the number of letters read correctly on the ETDRS chart by the study eye at 4 meters. ETDRS letters score could range from 0 to 100 letters at each assessment.
  A positive change from Baseline in ETDRS letter score indicated an improvement in visual acuity in the study eye. Change from Baseline calculated as observed post-baseline value - Baseline value.
Time Frame: Baseline and Weeks 4, 8, 16, 24, 32, 40, 48, and 52
Population: Full Analysis Set (Re-randomized): Consisted of all randomized participants, with treatment as the re-randomized treatment regardless of actual treatment received. Participants were included in the treatment group in which they were re-randomized. Analysis included participants with available data at Baseline and at each timepoint.
Measure: Mean (Standard Deviation); unit: Letters
Arm/Group | ABP 938 / ABP 938 | Aflibercept / Aflibercept | Aflibercept / ABP 938
Number analyzed (Participants) | 273 | 136 | 134
Letters
  Week 4: number analyzed (Participants) | 272 | 136 | 131
  Week 4 | 5.0 (6.57) | 5.4 (8.35) | 3.8 (8.19)
  Week 8: number analyzed (Participants) | 270 | 134 | 133
  Week 8 | 6.5 (8.10) | 7.6 (9.30) | 5.6 (8.86)
  Week 16 | 6.8 (8.69) | 7.5 (9.31) | 7.1 (9.32)
  Week 24: number analyzed (Participants) | 267 | 136 | 130
  Week 24 | 7.2 (9.63) | 7.1 (9.30) | 7.0 (10.12)
  Week 32: number analyzed (Participants) | 263 | 132 | 131
  Week 32 | 7.1 (11.00) | 8.7 (9.21) | 6.6 (11.11)
  Week 40: number analyzed (Participants) | 258 | 130 | 125
  Week 40 | 7.3 (11.00) | 8.1 (11.00) | 7.9 (10.08)
  Week 48: number analyzed (Participants) | 251 | 126 | 123
  Week 48 | 7.2 (11.51) | 8.7 (10.84) | 8.1 (10.74)
  Week 52: number analyzed (Participants) | 251 | 125 | 123
  Week 52 | 7.6 (11.60) | 9.4 (10.18) | 8.0 (11.14)
Statistical Analysis 1: Comparison: ABP 938 / ABP 938 vs Aflibercept / Aflibercept; Difference in mean change from Baseline at Week 4; Test type: Other; Difference between means = -0.1, 90% CI 2-sided [-1.3 to 1.2] — Estimated using ANCOVA model adjusted for the stratification factors geographic region (East Asia, Europe, North America) and Baseline BCVA as covariates
Statistical Analysis 2: Comparison: ABP 938 / ABP 938 vs Aflibercept / Aflibercept; Difference in mean change from Baseline at Week 8; Test type: Other; Difference between means = -0.8, 90% CI 2-sided [-2.3 to 0.7] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 3: Comparison: ABP 938 / ABP 938 vs Aflibercept / Aflibercept; Difference in mean change from Baseline at Week 16; Test type: Other; Difference between means = -0.3, 90% CI 2-sided [-1.9 to 1.2] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 4: Comparison: ABP 938 / ABP 938 vs Aflibercept / Aflibercept; Difference in mean change from Baseline at Week 24; Test type: Other; Difference between means = 0.4, 90% CI 2-sided [-1.3 to 2.1] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 5: Comparison: ABP 938 / ABP 938 vs Aflibercept / Aflibercept; Difference in mean change from Baseline at Week 32; Test type: Other; Difference between means = -1.3, 90% CI 2-sided [-3.1 to 0.5] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 6: Comparison: ABP 938 / ABP 938 vs Aflibercept / Aflibercept; Difference in mean change from Baseline at Week 40; Test type: Other; Difference between means = -0.5, 90% CI 2-sided [-2.3 to 1.4] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 7: Comparison: ABP 938 / ABP 938 vs Aflibercept / Aflibercept; Difference in mean change from Baseline at Week 48; Test type: Other; Difference between means = -1.2, 90% CI 2-sided [-3.2 to 0.8] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 8: Comparison: ABP 938 / ABP 938 vs Aflibercept / Aflibercept; Difference in mean change from Baseline at Week 52; Test type: Other; Difference between means = -1.5, 2% CI 2-sided [-3.4 to 0.5] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 9: Comparison: Aflibercept / Aflibercept vs Aflibercept / ABP 938; Difference in mean change from Baseline at Week 4; Test type: Other; Difference between means = -1.5, 90% CI 2-sided [-3.0 to 0.0] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 10: Comparison: Aflibercept / Aflibercept vs Aflibercept / ABP 938; Difference in mean change from Baseline at Week 8; Test type: Other; Difference between means = -1.9, 90% CI 2-sided [-3.6 to -0.2] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 11: Comparison: Aflibercept / Aflibercept vs Aflibercept / ABP 938; Difference in mean change from Baseline at Week 16; Test type: Other; Difference between means = -0.3, 90% CI 2-sided [-2.1 to 1.5] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 12: Comparison: Aflibercept / Aflibercept vs Aflibercept / ABP 938; Difference in mean change from Baseline at Week 24; Test type: Other; Difference between means = 0.0, 90% CI 2-sided [-1.9 to 2.0] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 13: Comparison: Aflibercept / Aflibercept vs Aflibercept / ABP 938; Difference in mean change from Baseline at Week 32; Test type: Other; Difference between means = -1.9, 90% CI 2-sided [-4.0 to 0.2] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 14: Comparison: Aflibercept / Aflibercept vs Aflibercept / ABP 938; Difference in mean change from Baseline at Week 40; Test type: Other; Difference between means = 0.0, 90% CI 2-sided [-2.2 to 2.2] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 15: Comparison: Aflibercept / Aflibercept vs Aflibercept / ABP 938; Difference in mean change from Baseline at Week 48; Test type: Other; Difference between means = -0.6, 90% CI 2-sided [-2.9 to 1.7] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 16: Comparison: Aflibercept / Aflibercept vs Aflibercept / ABP 938; Difference in mean change from Baseline at Week 52; Test type: Other; Difference between means = -1.2, 90% CI 2-sided [-3.5 to 1.1] — [estimate comment as in outcome 3, analysis 1]

4. Secondary Outcome: Percentage of Participants Who Gained at Least 10 Letters of Vision at Week 8
Description: Percentage of participants who gained at least 10 letters of vision was assessed based on the number of letters read correctly on the ETDRS chart by the study eye at 4 meters. ETDRS letters score could range from 0 to 100 letters at each assessment.
Time Frame: Week 8
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | ABP 938 | Aflibercept
Number analyzed (Participants) | 279 | 281
Percentage of participants | 29.4 [24.1 to 34.7] | 32.7 [27.3 to 38.2]
Statistical Analysis 1: Comparison: ABP 938 vs Aflibercept; Risk difference in percentage of participants who gained at least 10 letters of vision at Week 8; Test type: Other; Risk Difference (RD) = -3.4, 90% CI 2-sided [-9.8 to 3.1] — [estimate comment as in outcome 2, analysis 1]

5. Secondary Outcome: Percentage of Participants Who Gained at Least 15 Letters of Vision at Week 52
Description: Percentage of participants who gained at least 15 letters of vision was assessed based on the number of letters read correctly on the ETDRS chart by the study eye at 4 meters. ETDRS letters score could range from 0 to 100 letters at each assessment.
Time Frame: Week 52
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | ABP 938 / ABP 938 | Aflibercept / Aflibercept | Aflibercept / ABP 938
Number analyzed (Participants) | 251 | 125 | 123
Percentage of participants | 24.3 [19.0 to 29.6] | 29.6 [21.6 to 37.6] | 24.4 [16.8 to 32.0]
Statistical Analysis 1: Comparison: ABP 938 / ABP 938 vs Aflibercept / Aflibercept; Risk difference in percentage of participants who gained at least 15 letters of vision at Week 52; Test type: Other; Risk Difference (RD) = -5.3, 90% CI 2-sided [-13.6 to 2.5] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Aflibercept / Aflibercept vs Aflibercept / ABP 938; Risk difference in percentage of participants who gained at least 15 letters of vision at Week 52; Test type: Other; Risk Difference (RD) = -5.2, 90% CI 2-sided [-14.4 to 4.2] — [estimate comment as in outcome 2, analysis 1]

6. Secondary Outcome: Mean Change From Baseline in Choroidal Neovascularization (CNV) Area Size
Description: CNV area size was measured by fluorescein angiography.
  Change from Baseline calculated as observed post-baseline value - Baseline value.
Time Frame: Baseline and Weeks 8, 16, 24, and 52
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mm^2
Arm/Group | ABP 938 / ABP 938 | Aflibercept / Aflibercept | Aflibercept / ABP 938
Number analyzed (Participants) | 255 | 127 | 130
mm^2
  Week 8 | -4.962 (5.1604) | -5.479 (5.1023) | -5.169 (4.6943)
  Week 16: number analyzed (Participants) | 245 | 121 | 125
  Week 16 | -4.089 (5.3668) | -5.174 (5.2280) | -4.751 (4.8814)
  Week 24: number analyzed (Participants) | 242 | 119 | 118
  Week 24 | -4.323 (5.5972) | -5.308 (5.6238) | -5.121 (5.2776)
  Week 52: number analyzed (Participants) | 234 | 119 | 114
  Week 52 | -6.276 (6.2690) | -7.280 (5.8262) | -6.434 (5.2445)
Statistical Analysis 1: Comparison: ABP 938 / ABP 938 vs Aflibercept / Aflibercept; Difference in mean change from Baseline at Week 8; Test type: Other; Difference between means = -0.048, 90% CI 2-sided [-0.734 to 0.638] — Estimated using ANCOVA model with treatment, Baseline CNV measurement and the stratification factors geographic region (East Asia, Europe, North America) and Baseline BCVA (BCVA < 64 letters, BCVA ≥ 64 letters) as covariates
Statistical Analysis 2: Comparison: ABP 938 / ABP 938 vs Aflibercept / Aflibercept; Difference in mean change from Baseline at Week 16; Test type: Other; Difference between means = 0.431, 90% CI 2-sided [-0.367 to 1.229] — [estimate comment as in outcome 6, analysis 1]
Statistical Analysis 3: Comparison: ABP 938 / ABP 938 vs Aflibercept / Aflibercept; Difference in mean change from Baseline at Week 24; Test type: Other; Difference between means = 0.197, 90% CI 2-sided [-0.625 to 1.019] — [estimate comment as in outcome 6, analysis 1]
Statistical Analysis 4: Comparison: ABP 938 / ABP 938 vs Aflibercept / Aflibercept; Difference in mean change from Baseline at Week 52; Test type: Other; Difference between means = 0.156, 2% CI 2-sided [-0.561 to 0.872] — [estimate comment as in outcome 6, analysis 1]
Statistical Analysis 5: Comparison: Aflibercept / Aflibercept vs Aflibercept / ABP 938; Difference in mean change from Baseline at Week 8; Test type: Other; Difference between means = 0.105, 90% CI 2-sided [-0.682 to 0.891] — [estimate comment as in outcome 6, analysis 1]
Statistical Analysis 6: Comparison: Aflibercept / Aflibercept vs Aflibercept / ABP 938; Difference in mean change from Baseline at Week 16; Test type: Other; Difference between means = 0.245, 90% CI 2-sided [-0.667 to 1.158] — [estimate comment as in outcome 6, analysis 1]
Statistical Analysis 7: Comparison: Aflibercept / Aflibercept vs Aflibercept / ABP 938; Difference in mean change from Baseline at Week 24; Test type: Other; Difference between means = -0.116, 90% CI 2-sided [-1.065 to 0.834] — [estimate comment as in outcome 6, analysis 1]
Statistical Analysis 8: Comparison: Aflibercept / Aflibercept vs Aflibercept / ABP 938; Difference in mean change from Baseline at Week 52; Test type: Other; Difference between means = 0.647, 90% CI 2-sided [-0.186 to 1.479] — [estimate comment as in outcome 6, analysis 1]

7. Secondary Outcome: Mean Change From Baseline in Central Subfield Thickness (CST)
Description: CST was defined as the average thickness in the ETDRS central 1 mm diameter subfield (the central subfield) and was measured by spectral domain optical coherence tomography.
  Change from Baseline calculated as observed post-baseline value - Baseline value.
Time Frame: Baseline and Weeks 4, 8, 16, 24, 32, 40, 48, and 52
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: μm
Arm/Group | ABP 938 / ABP 938 | Aflibercept / Aflibercept | Aflibercept / ABP 938
Number analyzed (Participants) | 273 | 136 | 134
μm
  Week 4: number analyzed (Participants) | 270 | 136 | 131
  Week 4 | -136.5 (108.91) | -143.1 (107.32) | -149.7 (107.01)
  Week 8: number analyzed (Participants) | 269 | 134 | 132
  Week 8 | -145.9 (106.24) | -146.3 (110.39) | -167.4 (118.52)
  Week 16: number analyzed (Participants) | 273 | 135 | 134
  Week 16 | -125.2 (124.81) | -127.3 (103.35) | -143.2 (121.93)
  Week 24: number analyzed (Participants) | 265 | 133 | 128
  Week 24 | -130.8 (125.63) | -131.7 (102.98) | -151.2 (118.21)
  Week 32: number analyzed (Participants) | 262 | 132 | 131
  Week 32 | -133.2 (122.93) | -134.1 (116.02) | -154.8 (114.22)
  Week 40: number analyzed (Participants) | 257 | 130 | 124
  Week 40 | -132.3 (113.25) | -135.6 (119.07) | -155.7 (119.95)
  Week 48: number analyzed (Participants) | 251 | 125 | 123
  Week 48 | -132.3 (124.15) | -141.1 (112.29) | -157.8 (121.23)
  Week 52: number analyzed (Participants) | 250 | 125 | 123
  Week 52 | -157.1 (114.25) | -159.1 (108.82) | -177.4 (122.22)
Statistical Analysis 1: Comparison: ABP 938 / ABP 938 vs Aflibercept / Aflibercept; Difference in mean change from Baseline at Week 4; Test type: Other; Difference between means = 6.2, 90% CI 2-sided [-5.6 to 17.9] — Estimated using ANCOVA model with treatment, Baseline CST measurement and the stratification factors geographic region (East Asia, Europe, North America) and Baseline BCVA (BCVA < 64 letters, BCVA ≥ 64 letters) as covariates
Statistical Analysis 2: Comparison: ABP 938 / ABP 938 vs Aflibercept / Aflibercept; Difference in mean change from Baseline at Week 8; Test type: Other; Difference between means = 1.3, 90% CI 2-sided [-11.0 to 13.5] — [estimate comment as in outcome 7, analysis 1]
Statistical Analysis 3: Comparison: ABP 938 / ABP 938 vs Aflibercept / Aflibercept; Difference in mean change from Baseline at Week 16; Test type: Other; Difference between means = 1.9, 90% CI 2-sided [-12.9 to 16.6] — [estimate comment as in outcome 7, analysis 1]
Statistical Analysis 4: Comparison: ABP 938 / ABP 938 vs Aflibercept / Aflibercept; Difference in mean change from Baseline at Week 24; Test type: Other; Difference between means = 0.1, 90% CI 2-sided [-14.1 to 14.4] — [estimate comment as in outcome 7, analysis 1]
Statistical Analysis 5: Comparison: ABP 938 / ABP 938 vs Aflibercept / Aflibercept; Difference in mean change from Baseline at Week 32; Test type: Other; Difference between means = -1.2, 90% CI 2-sided [-15.3 to 12.9] — [estimate comment as in outcome 7, analysis 1]
Statistical Analysis 6: Comparison: ABP 938 / ABP 938 vs Aflibercept / Aflibercept; Difference in mean change from Baseline at Week 40; Test type: Other; Difference between means = 0.2, 90% CI 2-sided [-13.7 to 14.1] — [estimate comment as in outcome 7, analysis 1]
Statistical Analysis 7: Comparison: ABP 938 / ABP 938 vs Aflibercept / Aflibercept; Difference in mean change from Baseline at Week 48; Test type: Other; Difference between means = 7.0, 90% CI 2-sided [-7.4 to 21.4] — [estimate comment as in outcome 7, analysis 1]
Statistical Analysis 8: Comparison: ABP 938 / ABP 938 vs Aflibercept / Aflibercept; Difference in mean change from Baseline at Week 52; Test type: Other; Difference between means = 1.6, 2% CI 2-sided [-9.3 to 12.5] — [estimate comment as in outcome 7, analysis 1]
Statistical Analysis 9: Comparison: Aflibercept / Aflibercept vs Aflibercept / ABP 938; Difference in mean change from Baseline at Week 4; Test type: Other; Difference between means = 6.3, 90% CI 2-sided [-7.4 to 20.0] — [estimate comment as in outcome 7, analysis 1]
Statistical Analysis 10: Comparison: Aflibercept / Aflibercept vs Aflibercept / ABP 938; Difference in mean change from Baseline at Week 8; Test type: Other; Difference between means = -5.1, 90% CI 2-sided [-19.3 to 9.1] — [estimate comment as in outcome 7, analysis 1]
Statistical Analysis 11: Comparison: Aflibercept / Aflibercept vs Aflibercept / ABP 938; Difference in mean change from Baseline at Week 16; Test type: Other; Difference between means = -3.8, 90% CI 2-sided [-20.9 to 13.3] — [estimate comment as in outcome 7, analysis 1]
Statistical Analysis 12: Comparison: Aflibercept / Aflibercept vs Aflibercept / ABP 938; Difference in mean change from Baseline at Week 24; Test type: Other; Difference between means = -6.0, 90% CI 2-sided [-22.6 to 10.6] — [estimate comment as in outcome 7, analysis 1]
Statistical Analysis 13: Comparison: Aflibercept / Aflibercept vs Aflibercept / ABP 938; Difference in mean change from Baseline at Week 32; Test type: Other; Difference between means = -7.0, 90% CI 2-sided [-23.3 to 9.3] — [estimate comment as in outcome 7, analysis 1]
Statistical Analysis 14: Comparison: Aflibercept / Aflibercept vs Aflibercept / ABP 938; Difference in mean change from Baseline at Week 40; Test type: Other; Difference between means = -6.5, 90% CI 2-sided [-22.8 to 9.8] — [estimate comment as in outcome 7, analysis 1]
Statistical Analysis 15: Comparison: Aflibercept / Aflibercept vs Aflibercept / ABP 938; Difference in mean change from Baseline at Week 48; Test type: Other; Difference between means = -0.5, 90% CI 2-sided [-17.3 to 16.2] — [estimate comment as in outcome 7, analysis 1]
Statistical Analysis 16: Comparison: Aflibercept / Aflibercept vs Aflibercept / ABP 938; Difference in mean change from Baseline at Week 52; Test type: Other; Difference between means = 2.3, 90% CI 2-sided [-10.5 to 15.0] — [estimate comment as in outcome 7, analysis 1]

8. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a clinical trial participant. TEAEs were defined as those AEs that begin or increase in severity or frequency at or after the time of first treatment to the End of Study visit. Events of interest (EOIs) pre-specified for this study included endophthalmitis, retinal detachment, increase in intraocular pressure, and thromboembolic events. Serious AEs were defined as any untoward medical occurrence that meets at least 1 of the following serious criteria:
  * Results in death
  * Life-threatening
  * Requires inpatient hospitalization or prolongation of existing hospitalization
  * Results in persistent or significant disability/incapacity
  * Congenital anomaly/birth defect
  * Other medically important serious event.
Time Frame: Up to Week 52
Population: Safety Analysis Set: Consisted of all participants who received at least 1 dose of investigational product, with treatment assignment based on actual treatment received. TEAEs were collected for all participants who were re-randomized and received at least one dose of study drug post Week 16.
Measure: Count of Participants; unit: Participants
Groups:
- Through Week 16: ABP 938: Participants were treated with 2 mg (0.05 mL) of ABP 938 by IVT injection in the study eye every 4 weeks for the first 3 doses (i.e., Baseline/Day 1, Week 4, and Week 8).
- Through Week 16: Aflibercept: Participants were treated with 2 mg (0.05 mL) of aflibercept by IVT injection in the study eye every 4 weeks for the first 3 doses (i.e., Baseline/Day 1, Week 4, and Week 8).
- Post Week 16: ABP 938 / ABP 938: Participants who were initially treated with ABP 938 and remained on treatment with 2 mg (0.05 mL) of ABP 938 by IVT injection in the study eye every 8 weeks from Week 16 until Week 48.
- Post Week 16: Aflibercept / ABP 938: Participants who were initially treated with aflibercept and were re-randomized and treated with 2 mg (0.05 mL) of ABP-938 by IVT injection in the study eye every 8 weeks from Week 16 until Week 48.
- Post Week 16: Aflibercept / Aflibercept: Participants who were initially treated with aflibercept and were re-randomized and treated with 2 mg (0.05 mL) of aflibercept by IVT injection in the study eye every 8 weeks from Week 16 until Week 48.
Arm/Group | Through Week 16: ABP 938 | Through Week 16: Aflibercept | Post Week 16: ABP 938 / ABP 938 | Post Week 16: Aflibercept / ABP 938 | Post Week 16: Aflibercept / Aflibercept
Number analyzed (Participants) | 288 | 288 | 273 | 133 | 136
Participants
  Any TEAEs | 113 | 107 | 144 | 76 | 72
  Any EOIs | 6 | 3 | 9 | 8 | 2
  Any Serious TEAEs | 6 | 9 | 22 | 14 | 11

9. Secondary Outcome: Number of Participants Developing Binding Antidrug Antibodies (ADAs)
Description: Number of participants with positive post-baseline ADA result through Week 16 and post Week 16 with negative or no result at Baseline is reported.
Time Frame: Baseline up to Week 52
Population: Safety Analysis Set (Re-randomized and Treated): Consisted of all participants who received at least 1 dose of investigational product, with treatment assignment based on actual treatment received. Analysis included participants with available data at Baseline and at each timepoint.
Measure: Count of Participants; unit: Participants
Groups:
- Post Week 16: ABP 938 / ABP 938: Participants who were initially treated with 2 mg (0.05 mL) of aflibercept by IVT injection in the study eye every 4 weeks for the first 3 doses (i.e., Baseline/Day 1, Week 4, and Week 8) were re-randomized and treated with 2 mg (0.05 mL) of ABP 938 by IVT injection in the study eye every 8 weeks from Week 16 until Week 48.
Arm/Group | Through Week 16: ABP 938 | Through Week 16: Aflibercept | Post Week 16: ABP 938 / ABP 938 | Post Week 16: Aflibercept / ABP 938 | Post Week 16: Aflibercept / Aflibercept
Number analyzed (Participants) | 288 | 288 | 273 | 133 | 136
Participants | 1 | 4 | 4 | 3 | 0

ADVERSE EVENTS:
Time Frame: Up to Week 52
Description: All-cause mortality was collected for all participants enrolled/randomized in the study. Serious AEs and other AEs were collected for all participants who received at least one dose of study drug through Week 16. Serious AEs and other AEs were collected for all participants who were re-randomized and received at least one dose of study drug post Week 16.
Arm/Group | Through Week 16: ABP 938 | Through Week 16: Aflibercept | Post Week 16: ABP 938 / ABP 938 | Post Week 16: Aflibercept / ABP 938 | Post Week 16: Aflibercept / Aflibercept
All-Cause Mortality (participants affected / at risk) | 0/288 | 2/288 | 2/273 | 2/133 | 0/136
Serious Adverse Events (participants affected / at risk) | 6/288 | 9/288 | 22/273 | 14/133 | 11/136
Other Adverse Events (participants affected / at risk) | 18/288 | 15/288 | 20/273 | 17/133 | 17/136
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Through Week 16: ABP 938 (N=288) | Through Week 16: Aflibercept (N=288) | Post Week 16: ABP 938 / ABP 938 (N=273) | Post Week 16: Aflibercept / ABP 938 (N=133) | Post Week 16: Aflibercept / Aflibercept (N=136)
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Adrenal haematoma (Endocrine disorders) | 0 | 0 | 1 | 0 | 0
Retinal detachment (Eye disorders) | 0 | 0 | 1 | 0 | 0
Retinal haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 1
Visual acuity reduced (Eye disorders) | 0 | 0 | 0 | 0 | 1
Visual impairment (Eye disorders) | 0 | 0 | 0 | 0 | 1
Pneumatosis intestinalis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Cholangitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Arthropod-borne disease (Infections and infestations) | 0 | 0 | 0 | 0 | 1
COVID-19 (Infections and infestations) | 0 | 2 | 2 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 1 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 3 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Heart rate decreased (Investigations) | 0 | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0 | 0
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Invasive lobular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Rosai-Dorfman syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Transitional cell cancer of the renal pelvis and ureter (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 2 | 3 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Bladder neck obstruction (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0
Peripheral artery stenosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Subclavian artery stenosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Through Week 16: ABP 938 (N=288) | Through Week 16: Aflibercept (N=288) | Post Week 16: ABP 938 / ABP 938 (N=273) | Post Week 16: Aflibercept / ABP 938 (N=133) | Post Week 16: Aflibercept / Aflibercept (N=136)
Conjunctival haemorrhage (Eye disorders) | 12 | 11 | 4 | 8 | 8
Neovascular age-related macular degeneration (Eye disorders) | 6 | 4 | 16 | 10 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2022-05-16): https://cdn.clinicaltrials.gov/large-docs/47/NCT04270747/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-26): https://cdn.clinicaltrials.gov/large-docs/47/NCT04270747/SAP_001.pdf